CLINICAL TRIAL: NCT04333914
Title: A Prospective, Controlled, Randomized, Multicenter Study of the Efficacy of an Autophagy Inhibitor (GNS561), an Anti-NKG2A (Monalizumab) and an Anti-C5aR (Avdoralimab) Compared to the Standard of Care in Patients With Advanced or Metastatic Cancer and SARS-CoV-2 (COVID-19) Infection.
Brief Title: Prospective Study in Patients With Advanced or Metastatic Cancer and SARS-CoV-2 Infection
Acronym: IMMUNONCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET20-076 - IMMUNONCOVID-20; 2020-001373-70 (EudraCT Number)
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV-2 (COVID-19) Infection; Advanced or Metastatic Hematological or Solid Tumor
Keywords: Oncology; COVID-19; IL-6/IL-6 receptor pathway; Immunotherapy; GNS561; anti-C5aR; anti-NKG2A
MeSH Terms: conditions — COVID-19; Infections; Neoplasms | interventions — Standard of Care; avdoralimab; monalizumab

STUDY DESIGN:
Intervention Model Description: * COHORT 1 : Patients with mild symptoms or asymptomatic
  * COHORT 2 : Patients with moderate/severe symptoms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Autophagy inhibitor (GNS651) (Experimental)
  Interventions: Drug: Autophagy inhibitor (GNS651); Other: Standard of care
- Standard of care (Other)
  Interventions: Other: Standard of care
- anti-NKG2A (Monalizumab) (Experimental)
  Interventions: Other: Standard of care; Drug: Monalizumab
- anti-C5aR (Avdoralimab) (Experimental)
  Interventions: Other: Standard of care; Drug: Avdoralimab

INTERVENTIONS:
Drug: Autophagy inhibitor (GNS651) — Cohort 1 (arm B): 200mg q.d. orally for 10 consecutive days. If for any reason a treatment is not given within the allowed treatment window (± 12h) it will be cancelled (i.e., missed for that time point), and treatment will be resumed at the next dosing day.
  Arms: Autophagy inhibitor (GNS651)
Other: Standard of care — In cohorts 1 and 2, patients allocated in the standard of care arms should receive best supportive care, as per the investigator's discretion and the local routine practices. With regards to the respiratory symptoms and medical resoures at investigational site, the following should be given according to the patient's condition: oxygen supplementation, non-invasive ventilation, invasive ventilation, antibiotherapy, vasopressor support, renal replacement therapy, or extracorporeal membrane oxygenation.
  Additional care and medications should be administered in the patient's best interest.
Drug: Avdoralimab — Cohorte 2 (arm H): 500mg, intravenously, at Day 1 then 200mg once daily every 2 days during 14 Days
  Arms: anti-C5aR (Avdoralimab)
Drug: Monalizumab — Cohorte 2 (arm G) : 50mg (flat dose),intravenously, single infusion at Day 1.
  Arms: anti-NKG2A (Monalizumab)

SUMMARY:
A prospective, controlled, randomized, multicenter study whose goal is to compare the efficacy of an autophagy inhibitor (GNS561), an anti-NKG2A (monalizumab) and an anti-C5aR (avdoralimab) versus standard of care in patients with advanced or metastatic cancer who have Sars-CoV-2 infection not eligible to a resuscitation unit.

According to their severity level at the time of enrolment, eligible patients will be randomized into 2 different cohorts:

* COHORT 1 (mild symptoms or asymptomatic): GNS561 vs anti-NKG2A vs standard of care (randomization ratio 1:1:1).
* COHORT 2 (moderate/severe symptoms): anti-C5aR vs standard of care (randomization ratio 1:1).

ELIGIBILITY:
INCLUSION CRITERIA:

I1. Age 18 or older at the time of enrolment for women and age 60 or older at the time of enrolment for men.

I2. Histologically or cytologically confirmed diagnosis of advanced or metastatic hematological or solid tumor (hematological or solid tumor, any type and any localization).

I3. Documented diagnosis of COVID-19 (diagnostic test performed in a certified laboratory) without indication of transfer in a rescucitation unit.; Nota Bene : A maximum time of 7 days may have elapsed between the date of first symptoms and the date of consent for patient cohort 1 (mild). In cohort 2 (severe), up to 10 days may have elapsed since the first symptoms.

I4. Cohort 2: patients with pneumonia confirmed by chest imaging, and an oxygen saturation (Sao2) of 94% or less while they are breathing ambient air or a ratio of the partial pressure of oxygen (Pao2) to the fraction of inspired oxygen (Fio2) (Pao2:Fio2) at or below 300 mg Hg.

I5. Multidisciplinary approach that patient is not eligible for a transfer to Resuscitation Unit (either due to underlying medical condition - including cancer - or due to lack of available bed).

Note: Item cancelled (addendum 2 - October 2020)

I6. Life-expectancy longer than 3 months.

I7. Adequate bone marrow and end-organ function defined by the following laboratory results:

* Bone marrow:

  * Hemoglobin ≥ 9.0 g/dL,
  * Absolute Neutrophils Count (ANC) ≥ 1.0 Gi/L,
  * Platelets ≥ 100 Gi/L;
* Hepatic function:

  * Total serum bilirubin ≤ 1.5 x ULN (except patients with Gilbert's syndrome who must have total serum bilirubin ≤ 3.0 x ULN),
  * AST/ALT ≤ 5 ULN
* Renal function:

  * Serum creatinine ≤ 2.0 x ULN or Cr. Cl. ≥ 30ml/min/1.73m² (MDRD or CKD-EPI formula);

I8. Willingness and ability to comply with the study requirements;

I9. Signed and dated informed consent indicating that the patient has been informed of all the aspects of the trial prior to enrollment (in case of emergency situation, please refer to protocol section 12.1 PATIENT INFORMATION AND INFORMED CONSENT);

I10. Women of childbearing potential (Appendix 1) are required to have a negative serum pregnancy test within 72 hours prior to study treatment start. A positive urine test must be confirmed by a serum pregnancy test;

I11. Women of childbearing potential and male patients must agree to use adequate highly effective contraception (Appendix 1) for the duration of study participation and up to 6 months following completion of therapy;

I12. Patient must be covered by a medical insurance.

EXCLUSION CRITERIA:

E1. For cohort 1 only: Patient currently receiving therapy with an anti-NKG2A.

E2. For cohort 2 only: Patient currently receiving therapy with an anti-C5aR.

E3. Patient presents a contraindication to monalizumab treatment (cohort 1 only) or to avdoralimab (cohort 2 only) as per respective IB, including known hypersensitivity to one of these study drugs or severe hypersensitivity reaction to any monoclonal antibody.

E4. For cohort 1 only: Patient known to have intolerance or hypersensitivity to chloroquine or any quinoline derivatives (quinine, chloroquine, tafenoquine, hydroxychloroquine, mefloquine). Patients previously exposed to CQ, HCQ or other quinoline derivates should have interrupted their treatment at least 72h prior to randomization.

E5. Patient has active autoimmune disease that has required systemic treatment in the past 3 months before the date of randomisation or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids at doses higher than 10 mg/d prednisone equivalents or immunosuppressive agents.

Note 1: Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the study.

Note 2: Patients may received corticosteroids as required for the management of SARS-CoV-2-related symptoms.

E6. Patient requires the use of one of the following forbidden treatment during the study treatment period, including but not limited to :

* Major surgery
* Live vaccines. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever and BCG. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines, and are not allowed.

E7. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to the date of randomisation unstable arrhythmias or unstable angina, Known Left Ventricular Ejection Fraction (LVEF) < 50%.

Note: Patients with known coronary artery disease, congestive heart failure not meeting the above criteria must be on a stable medical regimen that is optimized in the opinion of the treating physician and in consultation with a cardiologist if appropriate.

E8. Patient has known active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening), known active hepatitis C (Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA at screening) or known Human Immunodeficiency Virus (HIV) infection (HIV 1/2 antibodies).

E9. Prior allogeneic bone marrow transplantation or solid organ transplant in the past.

E10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.

E11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

E12. Pregnant or breastfeeding patient, or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
28-day survival rate | 28 days from randomization
  28-day survival rate, defined by the proportion of patients still alive 28 days after randomization.
  If vital status at 28 days post randomisation is not available due to early transfer in an external resuscitation unit, patients will be considered as failure at the date of the transfer.
  Comparison of each experimental arm (GNS561 then monalizumab for cohort1 and avdoralimab for cohort2) to control arm will be performed using a Fisher exact test.

SECONDARY OUTCOMES:
Time to clinical improvement | 28 days from randomization
  Time to clinical improvement defined as the time from randomization to an improvement of two points (from the status at randomization) on a seven-category ordinal scale (WHO-ISARIC) or live discharge from the hospital, whichever comes first.
Clinical status | Day 7, Day 14, Day 28
  Clinical status will be assessed using a 7-point ordinal scale :
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO;
  7. Death.
Clinical status | Day 7, Day 14, Day 28
  The NEWS2 score (National Early Warning Score) allocates a score based on six physiological parameters (respiratory rate / oxygen saturation / systolic blood pressure / heart rate / consciousness / temperature).
  It Determines the degree of illness of a patient and prompts critical care intervention.
  The total possible score ranges from 0 to 21. The higher the score, the greater the clinical risk. A total score close to 0 corresponds to a low risk and a total score higher than 7 corresponds to a high risk.
Mean change in the ranking on the ordinal scale from baseline to D7, D14 and D28 | Day 7, Day 14, Day 28
  Mean change in clinical status from baseline will be assessed by using a 7-point ordinal scale.
Mean change in the ranking of the NEWS2 score from baseline to D7, D14 and D28 | Day 7, Day 14, Day 28
  Mean change in clinical status from baseline will be assessed by using the NEWS2 score (National Early Warning Score).
  The NEWS2 score (National Early Warning Score) allocates a score based on six physiological parameters (respiratory rate / oxygen saturation / systolic blood pressure / heart rate / consciousness / temperature).
  It Determines the degree of illness of a patient and prompts critical care intervention.
  The total possible score ranges from 0 to 21. The higher the score, the greater the clinical risk. A total score close to 0 corresponds to a low risk and a total score higher than 7 corresponds to a high risk.
Overall survival | 3 months (i.e. at the time of last patient last visit)
  Overall survival will be defined by the time from date of randomization until date of death, regardless of the cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Length of stay in Intensive Care Unit | 3 months (i.e. at the time of last patient last visit)
  The length of stay in Intensive Care Unit (from the date of admission in the Unit to the date of discharge).
Duration of mechanical ventilation or high flow oxygen devices | 3 months (i.e. at the time of last patient last visit)
  The duration of mechanical ventilation or high flow oxygen devices (from the date of intubation to the stop date of mechanical ventilation or high flow oxygen)
Duration of hospitalization | 3 months (i.e. at the time of last patient last visit)
  The duration of hospitalization (from the date of hospitalization to the date of definitive discharge for live patients)
Rate of throat swab negativation | Day 7, Day 14, Day 28
Quantitative SARS-CoV-2 virus in throat swab and blood samples | Day 7, Day 14, Day 28
The rate of secondary infection by other documented pathogens (bacteria, fungi) | Day 7, Day 14, Day 28 (if available)
Biological parameters | 3 months (i.e. at the time of last patient last visit)
  Changes from baseline in neutrophils count (G/L)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 months (i.e. at the time of last patient last visit)
  Treatment-Emergent Adverse Events, Serious Adverse Events, Suspected Unexpected Serious Adverse Reactions, New Safety Issues described using the NCI-CTC AE classification v5.
  Number of participants with a discontinuation or temporary suspension of study drugs (for any reason).
Cost-Effectiveness Analyses (CEA) | 3 months (i.e. at the time of last patient last visit)
  Incremental Cost-Effectiveness Ratios (ICERs) expressed in cost per Life Year Gained.
Biological parameters | 3 months (i.e. at the the time of last patient last visit)
  Changes from baseline in lymphocytes count (G/L)
Biological parameters | 3 months (i.e. at the the time of last patient last visit)
  Changes from baseline in platelets count (G/L)
Biological parameters | 3 months (i.e. at the the time of last patient last visit)
  Changes from baseline in hemoglobin count (g/dL)
Biological parameters | 3 months (i.e. at the the time of last patient last visit)
  Changes from baseline in CRP count (mg/L)
Biological parameters | 3 months (i.e. at the the time of last patient last visit)
  Changes from baseline in pro-inflammatory cytokine (IL6)
The rate of patients with SARS-CoV-2 IgG antibodies at D7, D14 and D28 | Day 7, Day 14, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Virginie AVRILLON, M.D., Principal Investigator — Centre Leon Berard; Jean-Yves BLAY, M.D., Ph.D., Principal Investigator — Centre Leon Berard
Locations (12):
- France (12):
  - Centre Léon Bérard, Lyon, Rhône
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - AP-HP Hôpital Saint Antoine, Paris
  - AP-HP La Pitié Salpétrière, Paris
  - Hôpital Saint-Joseph, Paris
  - AP-HP Tenon, Paris
  - AP-HP Hôpital Bichat Claude Bernard, Paris
  - GH Diaconesses Croix Saint Simon, Paris
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg
  - Institut Gustave Roussy, Villejuif